CLINICAL TRIAL: NCT03129789
Title: Volumetric Bladder Ultrasound Training for Pediatric Residents: Curriculum Implementation and Learning Trajectory
Brief Title: Volumetric Bladder Ultrasound Training for Pediatric Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Laura Watkins, Attending Physician, Northwell Health
Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 17-0032
Record Dates: First submitted 2017-04-14; First posted 2017-04-26 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Ultrasound Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants perform ultrasound and the principle investigator is unaware of the identity of the participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Volumetric Bladder Ultrasound Training — teaching residents to perform bladder volumetric ultrasound

SUMMARY:
Monitoring fluid balance is crucial in the care of critically ill children. There are several reasons urine output could be decreased. For example, the bladder could be empty because the patient isn't making urine due to dehydration, or the bladder could be full but the patient unable to urinate due to obstruction of the bladder outlet. It is prudent to distinguish this difference in the care of Pediatric Intensive Care Unit patients as the potential interventions vary and none is without potential drawbacks if used inappropriately. At present, there is no standard way to determine whether an oliguric patient has a bladder that is under- or over-filled. Bedside ultrasound is safe, non-invasive, painless, and relatively quick and can help assess bladder volume at the time of noted oliguria. Several studies in pediatrics endorse the use of ultrasound to approximately measure urine volume. Pediatric residents are frequently asked to manage patients' oliguria in the Pediatric Intensive Care Unit, however, they are not currently being trained how to use ultrasound to measure bladder volume. The investigators hypothesize that following a structured learning plan, by the end of their one-month Pediatric Intensive Care Unit rotations, pediatric residents will be able to independently and accurately measure bladder volume by ultrasound. Volumetric bladder ultrasound is an easily mastered bedside imaging technique. Its implementation could positively affect care of the critically ill infant or child.

ELIGIBILITY:
Inclusion Criteria:

* medical resident rotating through the Pediatric Intensive Care Unit

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
competency | 1 month
  participant correctly performs and accurately interprets bladder volume measurements as outlined above three consecutive times

SECONDARY OUTCOMES:
post-instruction questionnaire | 1 month
  assess knowledge of basic ultrasound image acquisition and interpretation, confidence in ability to use volumetric bladder ultrasound, satisfaction with attainment of a new skill, and critical evaluation of the curriculum
skill retention | 3 months
  test to determine if participants are able to correctly performs and accurately interprets bladder volume measurements 3 months after training

CONTACTS AND LOCATIONS:
Locations (1):
- Steven and Alexandra Cohen Childrens Medical Center of NY, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No